CLINICAL TRIAL: NCT07204353
Title: A Novel Surgical Procedure for Peri-implant Papilla Reconstruction in the Aesthetic Region: Modified Labial Pedicle Papilla Flap Technique With De-epithelialized Gingival Graft
Brief Title: Modified Labial Pedicle Papilla Flap (mLPPF) With or Without De-epithelialized Gingival Graft (dGG) for Peri-implant Papilla Reconstruction
Acronym: mLPPF-dGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cuneyt Asim Aral (Other)
Responsible Party: Sponsor-Investigator, Cuneyt Asim Aral, Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUCREC.2024.161
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: Peri-Implant Papilla Deficiency
Keywords: Peri-implant papilla reconstruction; Modified labial pedicle papilla flap (mLPPF); De-epithelialized gingival graft (dGG); Crestal mucosa thickness; Jemt papilla index; Dental implant esthetics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation. Papilla height, Jemt scores, and crestal mucosa thickness were measured using standardized intraoral photographs and STL files by independent examiners who were unaware of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Papilla-preserving incisions performed during implant uncovering, without additional flap modification or grafting.
  Interventions: Procedure: Papilla-preserving incision (Control)
- mLPPF group (Experimental): A modified labial pedicle papilla flap is advanced and sutured to reconstruct the peri-implant papilla, without connective tissue grafting.
  Interventions: Procedure: Modified Labial Pedicle Papilla Flap (mLPPF)
- mLPPF+dGG group (Experimental): A modified labial pedicle papilla flap is combined with placement of a de-epithelialized gingival graft harvested from the palate, sutured into the papillary region to enhance papilla reconstruction and increase mucosal thickness.
  Interventions: Procedure: Modified Labial Pedicle Papilla Flap with De-epithelialized Gingival Graft (mLPPF+dGG)

INTERVENTIONS:
Procedure: Papilla-preserving incision (Control) — Standard papilla-preserving incision without additional flap modification or connective tissue grafting. This group serves as the control, receiving only routine surgical access for implant site management.
  Arms: Control group
Procedure: Modified Labial Pedicle Papilla Flap (mLPPF) — Surgical reconstruction of the peri-implant papilla using the modified labial pedicle papilla flap technique. The flap is mobilized and sutured without adjunctive grafting procedures.
  Arms: mLPPF group
Procedure: Modified Labial Pedicle Papilla Flap with De-epithelialized Gingival Graft (mLPPF+dGG) — Surgical reconstruction of the peri-implant papilla combining the modified labial pedicle papilla flap with placement of a de-epithelialized gingival graft (dGG) at the papillary region to enhance soft tissue volume and stability.
  Arms: mLPPF+dGG group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of two surgical techniques for peri-implant papilla reconstruction in single-tooth implants in the maxillary anterior and premolar regions. A total of 80 cases with papilla deficiency were allocated into three groups: papilla-preserving incisions only (Control), modified labial pedicle papilla flap (mLPPF), and mLPPF combined with a de-epithelialized gingival graft (mLPPF+dGG). Clinical outcomes including papilla fill (Jemt scores), papilla height, and crestal mucosa thickness were assessed at baseline, immediately after surgery, two weeks postoperatively, and six months after final restoration. The primary goal is to determine whether combining connective tissue grafting with flap surgery provides superior and more stable papilla reconstruction compared with papilla preserving flap-only approaches.

DETAILED DESCRIPTION:
Peri-implant papilla deficiency remains one of the most challenging aspects of achieving esthetic success in implant dentistry, particularly in the anterior maxilla where soft tissue harmony plays a pivotal role. Despite the development of several surgical and prosthetic techniques, no universally accepted gold standard procedure or biomaterial has been established for papilla reconstruction.

This randomized controlled clinical trial was designed to investigate the clinical outcomes of two surgical approaches for peri-implant papilla reconstruction: the modified labial pedicle papilla flap (mLPPF) performed alone, and mLPPF combined with a de-epithelialized gingival graft (mLPPF+dGG). Patients presenting with single-tooth missing sites in the maxillary anterior or premolar regions, associated with papilla loss, were recruited. A total of 80 cases were allocated to three groups:

Control group - papilla-preserving incisions only,

mLPPF group - surgical papilla reconstruction with a modified pedicle flap,

mLPPF+dGG group - flap reconstruction combined with a connective tissue graft harvested and de-epithelialized from the palate.

Clinical outcomes included Jemt papilla index scores, papilla height (measured using standardized intraoral photography and STL files), and crestal mucosa thickness. Measurements were obtained at baseline (T0), immediately after surgery (T1), two weeks postoperatively (T2), and six months after prosthetic restoration (T3).

The primary hypothesis was that combining flap techniques with dGG would result in superior papilla fill and long-term tissue stability compared with flap-only or incision-only techniques. Statistical analyses confirmed that the mLPPF+dGG group demonstrated significantly higher Jemt scores, papilla height, and crestal mucosa thickness from the early postoperative period through the six-month follow-up. Moreover, strong positive correlations were identified between papilla height and crestal mucosa thickness, supporting the biological interplay between vertical mucosal thickness and papillary stability.

The trial provides randomized controlled evidence that the use of de-epithelialized gingival grafts in combination with pedicle flap surgery is a predictable and effective method for peri-implant papilla reconstruction, with potential implications for clinical practice in esthetically demanding cases.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for inclusion if they:

  * Were between 22 and 45 years of age
  * Voluntarily agreed to participate in the study
  * Had good periodontal health defined as full-mouth bleeding on probing scores, with <10%
  * Had a single missing tooth in the maxillary anterior or premolar region with both neighbouring teeth present
  * Had peri-implant papilla loss defined as JEMT score <3

Exclusion Criteria:

* Participants were excluded if they:

  * Were smokers
  * Had any systemic condition that could potentially influence study outcomes or implant success, such as diabetes mellitus, osteoporosis, or a history of radiotherapy
  * Were undergoing pharmacological treatment that could affect the results, including the use of bisphosphonates, immunosuppressive agents, or regular analgesic medications
  * Had clinical signs of peri-implant mucositis or peri-implantitis

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Papilla Height | Baseline (T0), İmmediatelly after surgery (T1), 2 weeks postoperatively (T2), and 6 months after final restoration (T3).
  Papilla height will be measured as the perpendicular distance from the papilla tip to a line connecting the zenith points of the two adjacent teeth, using standardized intraoral photographs and STL-based digital analysis.

SECONDARY OUTCOMES:
Change in Jemt Scores | Baseline (T0), 2 weeks postoperatively (T2), and 6 months after final restoration (T3).
  Jemt scores will be assessed based on the degree of papilla fill, ranging from 0 (no papilla) to 4 (hypertrophic papilla).
Change in Crestal Mucosa Thickness | Baseline (T0), 2 weeks postoperatively (T2), and 6 months after final restoration (T3).
  Crestal mucosa thickness will be measured at the mid-buccal aspect using a standardized endodontic reamer with silicone stopper under local anesthesia. Measurements will be confirmed through STL-based analysis.
Correlation Between Papilla Height and Crestal Mucosa Thickness | Baseline (T0), 2 weeks postoperatively (T2), and 6 months after final restoration (T3).
  The relationship between papilla height and crestal mucosa thickness will be analyzed to determine the impact of vertical soft tissue thickness on papilla stability.

CONTACTS AND LOCATIONS:
Overall Officials: Cüneyt A Aral, Study Chair — Inonu University
Locations (1):
- Inonu University Faculty of Dentistry, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choquet V, Hermans M, Adriaenssens P, Daelemans P, Tarnow DP, Malevez C. Clinical and radiographic evaluation of the papilla level adjacent to single-tooth dental implants. A retrospective study in the maxillary anterior region. J Periodontol. 2001 Oct;72(10):1364-71. doi: 10.1902/jop.2001.72.10.1364. PMID 11699478
- [Background] Gholami GA, Hariri S, Amid R, Roghanizadeh L, Kadkhodazadeh M, Mehdizadeh A, Youssefi N. Average and Maximum Papilla Heights around Dental Implants in the Anterior Maxillary Region: A Retrospective Clinical Study. Int J Dent. 2022 Feb 11;2022:4235946. doi: 10.1155/2022/4235946. eCollection 2022. PMID 35186085
- [Background] Tarnow DP, Magner AW, Fletcher P. The effect of the distance from the contact point to the crest of bone on the presence or absence of the interproximal dental papilla. J Periodontol. 1992 Dec;63(12):995-6. doi: 10.1902/jop.1992.63.12.995. PMID 1474471
- [Background] Botticelli D, Agabiti I, Yamada R, Maniwa N, Apaza Alccayhuaman KA, Nakajima Y. Identifying Key Factors in Papilla Growth Around Implants: Focus on Intraoral Negative Pressure. Dent J (Basel). 2025 Mar 13;13(3):124. doi: 10.3390/dj13030124. PMID 40136752
- [Background] Beagle JR. Surgical reconstruction of the interdental papilla: case report. Int J Periodontics Restorative Dent. 1992;12(2):145-51. PMID 1521996